CLINICAL TRIAL: NCT04966819
Title: Assessing Current Survivorship Care Needs of Rectal Cancer Patients and Piloting a Dedicated Survivorship Initiative
Brief Title: Rectal Cancer Shared Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Associate Professor, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-1995
Record Dates: First submitted 2021-07-05; First posted 2021-07-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Rectal Cancer; Low Anterior Resection Syndrome
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not possible to mask the participant nor the care provider. However, outcome assessor will be blinded to the treatment allocation when analyzing primary and secondary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survivorship Care (Experimental): Survivorship care will consist of:
  1. Regular meetings with the rectal cancer oncology pivot nurse
  2. Identification of a primary care physician
  3. Development of an individualized survivorship plan
  4. Educational resources for patients
  Interventions: Other: Survivorship Care Initiative
- Standard Care (No Intervention): The control arm will consist of patients treated at the same institution who are receiving standard of care. Standard of care consists of meeting with colorectal oncology pivot nurse as needed (i.e. by referral from specialist based on patient needs).

INTERVENTIONS:
Other: Survivorship Care Initiative — The survivorship initiative will consist of:
  (A) Regular meetings with the rectal cancer oncology pivot nurse (IPO). These meetings present an opportunity for patients to discuss any treatment-related distress or late and long-term side-effect.
  (B) Identification of a primary care physician. If the patient is not known to a Primary care physician (PCP), the IPO will add the patient to an accelerated waitlist.
  (C) Development of an individualized survivorship plan. During meetings with the oncology pivot nurse, a survivorship care plan will be populated, included information on patient risk factors, treatments completed, pathology findings, and future surveillance planned. This document will be reviewed by the treating colorectal surgeon, and will be subsequently shared with the oncology team, the PCP and the patient (if the patient desires).
  (D) Educational resources for patients. Patients will be offered educational materials to help address their specific needs.
  Arms: Survivorship Care

SUMMARY:
The investigators propose a multifaceted rectal cancer survivorship care program involving oncology specialists, nursing support and primary care physicians. This initiative centers on regular meetings with oncology nursing support, enhanced communication and coordination of care among clinicians including primary care physicians, and an educational platform for patients regarding the late and long-term effects of cancer. Initial efforts will target rectal cancer patients specifically as they have been identified as being at high risk of having unmet needs. Once we have realized measurable, successful implementation in this population, our hope is then to expand our initiative to all colon cancer patients.

DETAILED DESCRIPTION:
Rectal cancer is a life-altering diagnosis that can have long-lasting effects not only on one's physical health, but also their psychological, emotional and financial well-being. With advancements in both disease detection and therapeutic options, there is now a growing cohort of patients who have successfully completed active rectal cancer treatment and transitioned into post-treatment care. Unfortunately, the post-treatment phase has its own set of challenges. Lost in Transition was one of the first major publications to advocate for dedicated survivorship planning, raising awareness of the needs of cancer survivors. Since then, both the National Comprehensive Cancer Network (NCCN) and the American Cancer Society have released guidelines for survivorship care focused on prevention, surveillance, assessment, intervention, coordination of care and survivorship planning. Despite these efforts to bolster survivorship care, studies have found an average of 2.88 unmet needs among cancer survivors affecting physical, financial, educational, emotional and psychology domains. The investigators propose a multifaceted rectal cancer survivorship care program involving oncology specialists, nursing support and primary care physicians. This initiative centers on regular meetings with oncology nursing support, enhanced communication and coordination of care among clinicians including primary care physicians, and an educational platform for patients regarding the late and long-term effects of cancer. Initial efforts will target rectal cancer patients specifically as they have been identified as being at high risk of having unmet needs. Once the investigators have realized measurable, successful implementation in this population, the hope is then to expand this initiative to all colon cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years-old)
* rectal cancer patients who underwent curative intent treatment between 2019-2020 (i.e. in the last 2 years), including those who underwent surgical resection (abdominoperineal resection or restorative proctectomy with or without ileostomy) and those managed non-operatively, with chemoradiotherapy will be included.

Exclusion Criteria:

* Cannot be contacted by telephone
* Unable to read and comprehend English or French;
* Unable to give clear and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Short Form-Survivor Unmet Needs Survey (Unmet needs) at 12 months | 12 months after study start
  Score ranges from 0 to 4. Higher score means higher degree of unmet needs.

SECONDARY OUTCOMES:
National Comprehensive Cancer Network Distress Thermometer | Baseline, 3, 6, and 12 months after study start
  Score ranges from 0 (no distress) to 10 (extreme distress). Higher score means higher distress.
Global Quality of Life (QoL) | Baseline, 3, 6, and 12 months after study start
  Global QoL as measured by the European Organization for Research & Treatment of Cancer QoL questionnaire (EORTC QLQ-C30). Linear transformation is used to standardize raw score, so that scores range from 0 to 100; higher score represents better functioning or worse level of symptoms.
Short Form-Survivor Unmet Needs Survey (Unmet needs) | Baseline, 3, and 6 months after study start
  Score ranges from 0 to 4. Higher score means higher degree of unmet needs.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada